CLINICAL TRIAL: NCT00837486
Title: Reclaim Deep Brain Stimulation Clinical Study for Treatment-Resistant Depression
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: MedtronicNeuro (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 1626; G080033
Record Dates: First submitted 2009-02-03; First posted 2009-02-05 (Estimated); Results first posted 2015-05-28 (Estimated); Last update posted 2015-05-28 (Estimated); Status verified 2015-05

CONDITIONS: Depression
Keywords: Treatment Resistant Depression; Treatment Refractory Depression; Deep Brain Stimulation; Depression
MeSH Terms: conditions — Depression; Depressive Disorder, Treatment-Resistant

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Active Group - Active Stimulation (Active Comparator): Receive active stimulation with Reclaim™ DBS System
  Interventions: Device: Reclaim™ DBS System
- Control Group - Sham Stimulation (Sham Comparator): Receive sham stimulation with Reclaim™ DBS System
  Interventions: Device: Reclaim™ DBS System

INTERVENTIONS:
Device: Reclaim™ DBS System

SUMMARY:
Medtronic, Inc. sponsored an investigational study of the Reclaim™ Deep Brain Stimulation (DBS) System in people that have treatment-resistant depression. Depression is a mood disorder and a serious medical condition that affects millions of Americans. Depressive symptoms may include loss of interest in things typically enjoyed; decreased energy levels; difficulty concentrating or making decisions; restlessness; and feelings of pessimism, hopelessness, and worthlessness. Treatment-resistant depression is a chronic and severe form of depression characterized by failure to respond to traditional forms of treatment, such as antidepressant medications and electroconvulsive therapy. Treatment-resistant depression significantly impacts quality of life, productivity, and is a major contributor of disability world-wide.

This randomized, double-blind, sham stimulation-controlled, multi-center, prospective, parallel design study used deep brain stimulation technology to test whether active bilateral stimulation can safely and effectively improve depressive symptoms in patients with treatment-resistant depression compared to sham stimulation.

Participants meeting criteria for the study were implanted with the Reclaim DBS System. Participants in the active group, who received active stimulation, were compared to the control group, who received sham stimulation, during the 16-week blinded-treatment phase. All participants were monitored for changes in depressive symptoms. After the blinded-treatment phase, all participants received active stimulation.

Candidates for the trial were adults who had major depressive disorder and had not responded to several treatments for depression. Participants in the study continued to receive their current antidepressant medications while participating in the trial.

ELIGIBILITY:
Inclusion Criteria:

* Consent to participate in screening and study procedures by signing and dating the Informed Consent Form
* Are diagnosed with major depressive disorder (MDD)
* Have tried at least 4 different treatments, for example antidepressant medications, combinations of antidepressant medications, and/or electroconvulsive therapy (ECT)
* Screening MADRS score ≥ 28
* Have had the current major depressive episode persist for at least 2 years
* Females, if of child-bearing potential, must be using an acceptable method of birth control

Exclusion Criteria:

* Females: Currently pregnant
* Currently enrolled in or plan to enroll in any concurrent drug and/or device study that may confound the results of this study
* Have a neurological condition that may jeopardize the safety or the conduct of the study
* Have any medical conditions unsuitable for undergoing DBS surgery

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2009-02; Primary Completion 2010-12 (Actual); Study Completion 2013-04 (Actual)

CONTACTS AND LOCATIONS:
Locations (5):
- United States (5):
  - Massachusetts General Hospital, Charlestown, Massachusetts
  - Cleveland Clinic Foundation, Cleveland, Ohio
  - University of Pennsylvania, Philadelphia, Pennsylvania
  - University of Pittsburgh Medical Center, Pittsburgh, Pennsylvania
  - Butler Hospital, Providence, Rhode Island

REFERENCES:
- [Result] Dougherty DD, Rezai AR, Carpenter LL, Howland RH, Bhati MT, O'Reardon JP, Eskandar EN, Baltuch GH, Machado AD, Kondziolka D, Cusin C, Evans KC, Price LH, Jacobs K, Pandya M, Denko T, Tyrka AR, Brelje T, Deckersbach T, Kubu C, Malone DA Jr. A Randomized Sham-Controlled Trial of Deep Brain Stimulation of the Ventral Capsule/Ventral Striatum for Chronic Treatment-Resistant Depression. Biol Psychiatry. 2015 Aug 15;78(4):240-8. doi: 10.1016/j.biopsych.2014.11.023. Epub 2014 Dec 13. PMID 25726497
- [Derived] Giacomo ED, Placenti V, Colmegna F, Clerici M. Obsessive-Compulsive Disorder in Pregnancy and Postpartum: The Possible Etiologic Role and Implications of Obsessive-Compulsive Personality Disorder. J Clin Psychiatry. 2021 Oct 19;82(6):21lr14069. doi: 10.4088/JCP.21lr14069. No abstract available. PMID 34670028
- [Derived] Fairbrother N, Collardeau F. High Prevalence of Perinatal-Occurring Obsessive-Compulsive Disorder: Reply to Di Giacomo et al. J Clin Psychiatry. 2021 Oct 19;82(6):21lr14069a. doi: 10.4088/JCP.21lr14069a. No abstract available. PMID 34670027
- [Derived] Hitti FL, Cristancho MA, Yang AI, O'Reardon JP, Bhati MT, Baltuch GH. Deep Brain Stimulation of the Ventral Capsule/Ventral Striatum for Treatment-Resistant Depression: A Decade of Clinical Follow-Up. J Clin Psychiatry. 2021 Oct 19;82(6):21m13973. doi: 10.4088/JCP.21m13973. PMID 34670026
- [Derived] Kubu CS, Brelje T, Butters MA, Deckersbach T, Malloy P, Moberg P, Troster AI, Williamson E, Baltuch GH, Bhati MT, Carpenter LL, Dougherty DD, Howland RH, Rezai AR, Malone DA Jr. Cognitive outcome after ventral capsule/ventral striatum stimulation for treatment-resistant major depression. J Neurol Neurosurg Psychiatry. 2017 Mar;88(3):262-265. doi: 10.1136/jnnp-2016-313803. Epub 2016 Sep 22. PMID 27659923

RESULTS

PARTICIPANT FLOW:
Groups:
- Active Group-Active Stimulation: Receive active stimulation during the first 16 weeks after device implant.
- Control Group-Sham Stimulation: Receive sham stimulation during the first 16 weeks after device implant.
Period: Blinded-treatment Phase
Arm/Group | Active Group-Active Stimulation | Control Group-Sham Stimulation
Started | 16 | 14
Completed | 15 (One subject did not receive the allocated intervention.) | 14
Not Completed | 1 | 0
Not completed — Physician Decision | 1 | 0
Period: Long-term Follow-up Phase - Open Label
Arm/Group | Active Group-Active Stimulation | Control Group-Sham Stimulation
Started | 29 (All subjects received open-label stimulation during this phase.) | 0
Completed | 24 | 0
Not Completed | 5 | 0
Not completed — Physician Decision | 2 | 0
Not completed — Withdrawal by Subject | 2 | 0
Not completed — Death | 1 | 0

BASELINE CHARACTERISTICS:
Population: All enrolled participants are included.
Groups:
- Total: Total of all reporting groups
Arm/Group | Active Group-Active Stimulation | Control Group-Sham Stimulation | Total
Number analyzed (Participants) | 16 | 14 | 30
Age, Continuous [Mean (Standard Deviation); unit: years] | 46.6 (14.4) | 48.9 (8.9) | 47.7 (12.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8 | 5 | 13
  Male | 8 | 9 | 17
Region of Enrollment [Number; unit: participants]
  United States | 16 | 14 | 30
Baseline depression score [Mean (Standard Deviation); unit: units on a scale] — Montgomery-Åsberg Depression Rating Scale (MADRS); total score can range from 0 (no symptoms) to 60 (severe depression)
  units on a scale | 37.0 (5.1) | 36.4 (3.3) | 36.7 (4.3)

OUTCOME MEASURES:

1. Primary Outcome: Responders
Description: Montgomery-Åsberg Depression Rating Scale (MADRS); total score can range from 0 (no symptoms) to 60 (severe depression). Response is defined as at least a 50% improvement (decline) in MADRS score. Responder rate is the proportion of participants who experience response.
Time Frame: Baseline to 16 weeks
Population: 29 of the 30 subjects are included in this analysis. One active group subject did not receive the allocated treatment, and is not included in the primary and secondary efficacy outcome analyses.
Measure: Number; unit: participants
Arm/Group | Active Group-Active Stimulation | Control Group-Sham Stimulation
Number analyzed (Participants) | 15 | 14
participants | 3 | 2
Statistical Analysis 1: Comparison: Active Group-Active Stimulation vs Control Group-Sham Stimulation; The study originally required a sample size of 208 subjects in order to have 90% power to detect a statistically significant difference between the responder rate of the active and control groups. With this 30-subject cohort, and only 29 subjects completing the blinded-treatment phase per protocol, the comparison of response rates was not adequately powered. The P-value is presented only to describe the outcomes of the two groups; Test type: Superiority or Other; p = 0.53, Fisher Exact — one-sided P-value per protocol responder rates: Active Group = 20.0%, Control Group = 14.3%

2. Secondary Outcome: Depression Change
Description: Montgomery-Åsberg Depression Rating Scale (MADRS); total score can range from 0 (no symptoms) to 60 (severe depression). Improvement is measured by the groups' mean percent change in MADRS score. An improvement is represented by a decline in MADRS (a negative percent change).
Time Frame: Baseline to 16 weeks
Population: One active group subject did not receive the allocated treatment, and is not included in the primary and secondary efficacy outcome analyses.
Measure: Mean (Standard Deviation); unit: percentage change from baseline
Arm/Group | Active Group-Active Stimulation | Control Group-Sham Stimulation
Number analyzed (Participants) | 15 | 14
percentage change from baseline | -19.6 (34.9) | -24.6 (28.8)

3. Secondary Outcome: Quality of Life Change
Description: Quality of Life Enjoyment and Satisfaction Questionnaire Short Form (Q-LES-Q-SF); total score can range from 0 to 100 with higher scores indicating a better quality of life. Improvement is measured by the groups' mean change in Q-LES-Q-SF score. An improvement is represented by an increase in Q-LES-Q-SF (a positive change).
Time Frame: Baseline to 16 weeks
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: change from baseline score
Arm/Group | Active Group-Active Stimulation | Control Group-Sham Stimulation
Number analyzed (Participants) | 15 | 14
change from baseline score | 10.2 (24.8) | 9.8 (18.8)

4. Other Pre Specified Outcome: Long-term Open-label Responders
Description: This measure is for long-term, open-label stimulation. Response is defined as at least a 50% improvement (decline) in MADRS score. Responder rate is the proportion of participants who experience response. All enrolled participants are included in the analysis, even if they withdrew early. Participants that withdrew early are counted as non-responders.
Time Frame: at the 24-month visit
Population: 29 participants started the the Long-Term Follow-up Phase and 24 completed the phase, but all 30 enrolled participants are included in the analysis. Participants that withdrew early are counted as non-responders.
Measure: Number; unit: participants
Groups:
- Long-term Open-label Treatment: All subjects received open-label active stimulation after the 16 week blinded-treatment phase.
Arm/Group | Long-term Open-label Treatment
Number analyzed (Participants) | 30
participants | 7

5. Other Pre Specified Outcome: Therapy-related Adverse Events
Description: Adverse events related to the device, implant procedure, and/or stimulation are reported. Events with a prevalence of greater than 5% of subjects are reported. This measure describes the experience of all study participants (both Active and Control Groups combined), and includes the operative, blinded-treatment,and the long-term open-label follow-up phases combined. Active Group participants began therapy after randomization, while Control Group participants began therapy after 16 weeks of sham stimulation.
Time Frame: from enrollment to study closure (average follow-up of 36 months)
Population: All enrolled participants are included in the analysis.
Measure: Number; unit: participants
Groups:
- All Enrolled Subjects: The 30 subjects were followed an average of 36 months after enrollment.
Arm/Group | All Enrolled Subjects
Number analyzed (Participants) | 30
participants
  Device - Implant site pain | 7
  Device - Paraesthesia | 4
  Procedure - Implant site pain | 8
  Procedure - Implant site infection | 5
  Procedure - Dermatitis contact | 2
  Procedure - Face oedema | 2
  Procedure - Headache | 2
  Procedure - Hypersensitivity | 2
  Stimulation - Insomnia | 15
  Stimulation - Depression | 8
  Stimulation - Hypomania | 8
  Stimulation - Irritability | 8
  Stimulation - Anxiety | 7
  Stimulation - Fatigue | 6
  Stimulation - Headache | 6
  Stimulation - Agitation | 5
  Stimulation - Sleep disorder | 5
  Stimulation - Disturbance in attention | 4
  Stimulation - Suicidal ideation | 4
  Stimulation - Disinhibition | 3
  Stimulation - Memory impairment | 3
  Stimulation - Paraesthesia | 3
  Stimulation - Energy increased | 2
  Stimulation - Impulsive behaviour | 2
  Stimulation - Nausea | 2
  Stimulation - Thinking abnormal | 2
  Stimulation - Weight increased | 2

ADVERSE EVENTS:
Time Frame: 16 weeks
Description: Adverse event results for the blinded-treatment phase only. All randomized subjects were included in adverse event summaries.
Arm/Group | Active Group-Active Stimulation | Control Group-Sham Stimulation
Serious Adverse Events (participants affected / at risk) | 4/16 | 4/14
Other Adverse Events (participants affected / at risk) | 15/16 | 14/14
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Active Group-Active Stimulation (N=16) | Control Group-Sham Stimulation (N=14)
Depression (Psychiatric disorders) | 1 | 3
Suicidal ideation (Psychiatric disorders) | 1 | 0
Disinhibition (Psychiatric disorders) | 1 | 0
Femoral arterial stenosis (Vascular disorders) | 1 | 0
Wound infection staphylococcal (Infections and infestations) | 0 | 1
Neurostimulator protrusion (Injury, poisoning and procedural complications) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Active Group-Active Stimulation (N=16) | Control Group-Sham Stimulation (N=14)
Implant site pain (General disorders) | 4 | 2
Depression (Psychiatric disorders) | 4 | 0
Insomnia (Psychiatric disorders) | 4 | 3
Fall (Injury, poisoning and procedural complications) | 1 | 3
Fatigue (General disorders) | 3 | 0
Hypertension (Vascular disorders) | 3 | 0
Irritability (Psychiatric disorders) | 3 | 0
Suicidal ideation (Psychiatric disorders) | 1 | 0
Headache (Nervous system disorders) | 2 | 1
Influenza (Infections and infestations) | 1 | 1
Disinhibition (Psychiatric disorders) | 1 | 0
Hypomania (Psychiatric disorders) | 2 | 0
Upper respiratory tract infection (Infections and infestations) | 2 | 0
Drug withdrawal syndrome (General disorders) | 1 | 1
Gastroenteritis viral (Infections and infestations) | 1 | 1
Sleep disorder (Psychiatric disorders) | 1 | 1
Tremor (Nervous system disorders) | 1 | 1
Localised infection (Infections and infestations) | 0 | 2
Abdominal pain (Gastrointestinal disorders) | 1 | 0
Adnexa uteri mass (Reproductive system and breast disorders) | 1 | 0
Bunion (Musculoskeletal and connective tissue disorders) | 1 | 0
Cognitive disorder (Nervous system disorders) | 1 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Dysphagia (Gastrointestinal disorders) | 1 | 0
Energy increased (General disorders) | 1 | 0
Eye pain (Eye disorders) | 1 | 0
Hypersomnia (Nervous system disorders) | 1 | 0
Hyporeflexia (Nervous system disorders) | 1 | 0
Mania (Psychiatric disorders) | 1 | 0
Neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Ocular hyperaemia (Eye disorders) | 1 | 0
Sinus congestion (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Somnolence (Nervous system disorders) | 1 | 0
Toothache (Gastrointestinal disorders) | 1 | 0
Transient ischaemic attack (Nervous system disorders) | 1 | 0
Allodynia (General disorders) | 0 | 1
Animal bite (Injury, poisoning and procedural complications) | 0 | 1
Back injury (Injury, poisoning and procedural complications) | 0 | 1
Balance disorder (Nervous system disorders) | 0 | 1
Bursitis (Musculoskeletal and connective tissue disorders) | 0 | 1
Constipation (Gastrointestinal disorders) | 0 | 1
Early morning awakening (Psychiatric disorders) | 0 | 1
Fungal infection (Infections and infestations) | 0 | 1
Menstruation irregular (Reproductive system and breast disorders) | 0 | 1
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 | 1
Nasopharyngitis (Infections and infestations) | 0 | 1
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 | 1
Paraesthesia (Nervous system disorders) | 0 | 1
Purging (Psychiatric disorders) | 0 | 1
Restless legs syndrome (Nervous system disorders) | 0 | 1
Rotator cuff syndrome (Musculoskeletal and connective tissue disorders) | 0 | 1
Tinnitus (Ear and labyrinth disorders) | 0 | 1
Upper respiratory tract congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 1

LIMITATIONS AND CAVEATS:
With this 30-subject cohort, and only 29 subjects completing the blinded-treatment phase per protocol, the comparisons of response rates and improvements were not adequately powered.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The disclosure restrictions on the PI allow for the sponsor to review results communications prior to public release and to embargo communications regarding trial results for a period that is less than or equal to 90 days from the time submitted to sponsor for review. The sponsor is also allowed to require changes for technical correctness and to protect confidential information, copyrightable or patentable material; and when reasonably requested, extend the embargo up to an additional 90 days.